CLINICAL TRIAL: NCT02621411
Title: Preoperative Screen for Substance Abuse in Trauma Patients Undergoing Emergency Operation: a Prospective Observational Study
Brief Title: Observational Study of Preoperative Screen for Substance Abuse
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Doctor, Associate professor, West China Hospital
Other Study IDs: WCH2015-100
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Preoperative Screen for Substance Abuse in in Patients Undergoing Emergency Operation
Keywords: Substance abuse; Emergency operation; Preoperative screen
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Substance abuser group: After preoperative screen by application of ICG test cassette, this group of patients are found current use of the certain substance(s).
  Interventions: Drug: Substance use
- Non-substance abuser group: After preoperative screen by application of ICG test cassette, this group of patients are not found use of any substance.

INTERVENTIONS:
Drug: Substance use — Patients are found use of substances by preoperative screen
  Groups: Substance abuser group

SUMMARY:
Substance abuse is a growing problem world wide, and treatment of substance abusers in the perioperative period, especially for emergency operation is challenging. The objectives of this study are to determine the proportions of substance abusers in the trauma patients undergoing emergency operation by preoperative screen, observe the differences of consumption of anesthetics and other medications during perioperative period between substance abusers and non-abusers, as well as postoperative complications, and explore an optimal scheme for substance abusers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16~70 years；
* Informed consent signed

Exclusion Criteria:

* Aged<16 years or >70 years；
* Refuse to sign consent;
* Other conditions that may preclude the patients from the study, such as language barrier, psychiatric disorders, unable to attend research center for follow up.
* Patients who enrolled to another research study or are taking experimental medication in last 3 months prior to this study.
* Not suitable for the study, after assessment by the investigators.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The trauma patients undergoing emergency operation
Sampling Method: Probability Sample
Enrollment: 1031 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion of substance abuser in all the emergency operation patients | 1 year
  The proportion will be calculated as the number of substance abusers / total number of enrolled calculated as the number of substance abusers / total number of enrolled patients

SECONDARY OUTCOMES:
Perioperative consumption of medications | 1 day
  Perioperative consumption of sulfentanil, midazolam, propofol, and muscle relaxant in substance abusers and non-abusers.
Incidence and severity of postoperative complications | 30 days

OTHER OUTCOMES:
Proportion of HIV, HCV, syphilis positive in substance abusers and non-abusers. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Study Director — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China